CLINICAL TRIAL: NCT01672866
Title: A Phase 2b, Dose-Ranging, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of GS-6624, a Monoclonal Antibody Against Lysyl Oxidase-Like Molecule 2 (LOXL2), in Subjects With Advanced Liver Fibrosis But Not Cirrhosis Secondary to Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Safety and Efficacy of Simtuzumab (SIM, GS-6624) in Adults With Advanced Liver Fibrosis But Not Cirrhosis Secondary to Non-Alcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-321-0105; 2012-002488-88 (EudraCT Number)
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Liver Fibrosis Due to NASH
Keywords: NASH; noncirrhotic; Monoclonal antibody; LOXL2; Simtuzumab; Nonalcoholic Steatohepatitis; NAFLD; Liver biopsy; MRE; Liver fibrosis; Ishak
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — simtuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SIM 75 mg (Experimental): During the Randomized Double-Blind Phase, participants will receive SIM 75 mg via subcutaneous injection once weekly for up to 240 weeks. During the optional Open-Label Phase, participants will receive SIM 125 mg via subcutaneous injection once weekly for up to an additional 240 weeks.
  Interventions: Biological: SIM
- SIM 125 mg (Experimental): During the Randomized Double-Blind Phase, participants will receive SIM 125 mg via subcutaneous injection once weekly for up to 240 weeks. During the optional Open-Label Phase, participants will receive SIM 125 mg via subcutaneous injection once weekly for up to an additional 240 weeks.
  Interventions: Biological: SIM
- Placebo (Placebo Comparator): During the Randomized Double-Blind Phase, participants will receive placebo to match SIM via subcutaneous injection once weekly for up to 240 weeks. During the optional Open-Label Phase, participants will receive SIM 125 mg via subcutaneous injection once weekly for up to an additional 240 weeks.
  Interventions: Biological: Placebo; Biological: SIM

INTERVENTIONS:
Biological: Placebo — Placebo to match SIM via subcutaneous injection every week
  Arms: Placebo
Biological: SIM — Subcutaneous injection every week
  Other Names: GS-6624

SUMMARY:
The primary objective of this study is to evaluate whether SIM (formerly referred to as GS-6624) is effective at preventing the histologic progression of liver fibrosis and the clinical progression to cirrhosis in participants with NASH.

It will consist of 2 phases:

* Randomized Double-Blind Phase
* Open-Label Phase (optional)

ELIGIBILITY:
Key Inclusion Criteria:

* Adults with chronic liver disease due to NASH defined as macrovesicular steatosis involving > 5% of hepatocytes on a liver biopsy with associated lobular inflammation
* Stage 3-4 fibrosis by Ishak score on a liver biopsy
* Exclusion of other causes of liver disease including viral hepatitis and alcoholic liver disease
* Must have aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 10 x Central Laboratory Upper Limit of Normal (clULN)
* Must have serum creatinine < 2.0 mg/dL
* A negative serum pregnancy test is required for females of childbearing potential
* All sexually active females of childbearing potential must agree to use a protocol recommended method of contraception during intercourse throughout the study and for 90 days following the last dose of study medication
* Lactating females must agree to discontinue nursing before starting study treatment
* Males, if not vasectomized, are required to use barrier contraception (condom plus spermicide) during heterosexual intercourse from the screening through the study completion and for 90 days following the last dose of study drug.

Key Exclusion Criteria:

* Pregnant or breast feeding
* Cirrhosis of the liver
* Any history of hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding
* Weight reduction surgery in the past 5 years
* Positive for hepatitis C virus (HCV) RNA
* Positive for HBsAg
* Alcohol consumption greater than 21oz/week for males or 14oz/week for females
* Positive urine screen for amphetamines, cocaine or opiates (i.e. heroin, morphine) at screening.
* Clinically significant cardiac disease
* History of malignancy, other than non-melanomatous skin cancer, within 5 years prior to screening
* Major surgical procedure within 30 days prior to screening or the presence of an open wound
* Known hypersensitivity to the investigation product or any of its formulation excipients
* History of bleeding diathesis within 6 months of screening
* Unavailable for follow-up assessment or concern for individual's compliance with the protocol procedures;
* Participation in an investigational trial of a drug or device within 30 days prior to screening
* BMI < 18 kg/m^2

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (68):
- United States (41):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Southern California Liver Centers, Coronado, California
  - University of California, San Diego (UCSD), San Diego, California
  - University of California San Francisco (UCSF), San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Miami Veterans Administration Healthcare System, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnnesota Gastroenterology, PA, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis University Hospital, St Louis, Missouri
  - State University Of New York, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Liver Institute of Virginia, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bucheon St. Marys Hospital, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Belgium (3):
  - Hôpital Erasme, Brussels
  - Université Catholique de Louvain, Brussels
  - UZ Ghent, Ghent
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - London Health Science Center, London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- France (4):
  - Hopital Beaujon, Clichy
  - Hospital Saint-Antoine, Paris
  - Groupe Hospitalier Pitié- Salpétrière, Paris
  - CHU Strasbourg Hôpital Civil, Strasbourg
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterologisch-Hepatologisches Zentrum Kiel, Kiel
  - EUGASTRO GmbH, Leipzig
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Modena Policlinico, Modena
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Fundacion De Investigacion, San Juan, Puerto Rico
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario Puerta de Hierro, Majadahonda
- United Kingdom (5):
  - John Radcliffe Hospital, Headington
  - The Royal London Hospital, London
  - Royal Free Hospital, Pond Street, London
  - King's College Hospital NHS Foundation Trust No. 1 Account, London
  - Nottingham University Hospitals Queens Medica, Nottingham

REFERENCES:
- [Result] Sanyal A, Harrison S, Ratziu V, Abdelmalek M, Diehl A, Caldwell S, et al. Changes in fibrosis, but not the NAFLD Activity Score (NAS), are associated with disease progression in patients with nonalcoholic steatohepatitis (NASH) and advanced fibrosis. J Hepatol 2017; 66 (1): S2.
- [Result] Sanyal A, Abdelmalek M, Diehl A, Caldwell S, Shiffman M, Ghalib R, et al. Efficacy and safety of simtuzumab for the treatment of nonalcoholic steatohepatitis with bridging fibrosis or cirrhosis: results of two phase 2b, dose-ranging, randomized, placebo-controlled trials. J Hepatol 2017; 66 (1): S54.
- [Result] Ratziu V, Sanyal A, Torres D, Hinrichsen H, Serfaty L, Bambha K, et al. Impact of weight reduction on serum markers and liver histology including progression to cirrhosis in patients with nonalcoholic steatohepatitis (NASH) and bridging fibrosis. J Hepatol 2017; 66 (1): S594.
- [Result] Shea PR, Sanyal A, Harrison S, Ratziu V, Loomba R, Caldwell S, et al. PNPLA3 variants confer an increased risk of advanced fibrosis due to non-alcoholic steatohepatitis. J Hepatol 2016; 64 (2): S493.
- [Result] Shea PR, Sanyal A, Rockey DC, Loomba R, Diehl AM, Kleinstein SE, et al. Genome-wide association study of clinically significant portal hypertension in patients with nonalcoholic steatohepatitis and advanced fibrosis. J Hepatol 2016; 64 (2): S280.
- [Result] Goodman ZD, Alaparthi L, Monge F, Patel K, Loomba R, Caldwell SH, et al. Correlations between hepatic morphometric collagen content, histologic fibrosis staging, and serum markers in patients with advanced fibrosis due to nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 906A.
- [Result] Harrison SA, Goodman ZD, Ratziu V, Loomba R, Diehl AM, Lawitz E, et al. Serum lysyl oxidase-like-2 (sLOXL2) levels correlate with fibrosis stage in patients with nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 910A.
- [Result] Ratziu V, Sanyal AJ, Loomba R, Caldwell SH, Ghalib RH, Torres DM, et al. Characterization of insulin resistance in patients with advanced fibrosis due to nonalcoholic steatohepatitis (NASH). Hepatol 2015; 62 (1): 1298A-1299A.
- [Derived] Loomba R, Huang DQ, Sanyal AJ, Anstee QM, Trauner M, Lawitz EJ, Ding D, Ma L, Jia C, Billin A, Huss RS, Chung C, Goodman Z, Wong VW, Okanoue T, Romero-Gomez M, Abdelmalek MF, Muir A, Afdhal N, Bosch J, Harrison S, Younossi ZM, Myers RP. Liver stiffness thresholds to predict disease progression and clinical outcomes in bridging fibrosis and cirrhosis. Gut. 2023 Mar;72(3):581-589. doi: 10.1136/gutjnl-2022-327777. Epub 2022 Sep 9. PMID 36750244
- [Derived] Younossi ZM, Anstee QM, Wai-Sun Wong V, Trauner M, Lawitz EJ, Harrison SA, Camargo M, Kersey K, Subramanian GM, Myers RP, Stepanova M. The Association of Histologic and Noninvasive Tests With Adverse Clinical and Patient-Reported Outcomes in Patients With Advanced Fibrosis Due to Nonalcoholic Steatohepatitis. Gastroenterology. 2021 Apr;160(5):1608-1619.e13. doi: 10.1053/j.gastro.2020.12.003. Epub 2020 Dec 8. PMID 33307033
- [Derived] Harrison SA, Abdelmalek MF, Caldwell S, Shiffman ML, Diehl AM, Ghalib R, Lawitz EJ, Rockey DC, Schall RA, Jia C, McColgan BJ, McHutchison JG, Subramanian GM, Myers RP, Younossi Z, Ratziu V, Muir AJ, Afdhal NH, Goodman Z, Bosch J, Sanyal AJ; GS-US-321-0105 and GS-US-321-0106 Investigators. Simtuzumab Is Ineffective for Patients With Bridging Fibrosis or Compensated Cirrhosis Caused by Nonalcoholic Steatohepatitis. Gastroenterology. 2018 Oct;155(4):1140-1153. doi: 10.1053/j.gastro.2018.07.006. Epub 2018 Jul 7. PMID 29990488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and North America. The first participant was screened on 05 December 2012. The last study visit occurred on 29 December 2016.
Pre-assignment Details: 631 participants were screened.
Groups:
- SIM 75 mg: Blinded Phase: Participants received simtuzumab (SIM) 75 mg via subcutaneous injection weekly for up to 240 weeks. Open-Label Phase: Participants received SIM 125 mg via subcutaneous injection weekly for up to an additional 240 weeks.
- SIM 125 mg: Blinded Phase: Participants received SIM 125 mg via subcutaneous injection weekly for up to 240 weeks. Open-Label Phase: Participants received SIM 125 mg via subcutaneous injection weekly for up to an additional 240 weeks.
- Placebo: Blinded Phase: Participants received placebo to match SIM via subcutaneous injection weekly for up to 240 weeks. Open-Label Phase: Participants received SIM 125 mg via subcutaneous injection weekly for up to an additional 240 weeks.
Period: Blinded Phase (up to 240 Weeks)
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Started | 74 | 74 | 74
Completed | 0 | 0 | 0
Not Completed | 74 | 74 | 74
Not completed — Study Terminated by Sponsor | 40 | 42 | 35
Not completed — Withdrew Consent | 9 | 8 | 12
Not completed — Lost to Follow-up | 3 | 3 | 5
Not completed — Adverse Event | 3 | 3 | 3
Not completed — Investigator's Discretion | 3 | 3 | 2
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Randomized but Never Treated | 3 | 0 | 0
Not completed — Met protocol-specified reason(s) | 11 | 15 | 16
Period: Open-Label Phase (up to 240 Weeks)
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Started | 11 (Met protocol-specified reason(s) for study discontinuation during Blinded Phase & entered Open-Label) | 15 (Met protocol-specified reason(s) for study discontinuation during Blinded Phase & entered Open-Label) | 16 (Met protocol-specified reason(s) for study discontinuation during Blinded Phase & entered Open-Label)
Completed | 0 | 0 | 0
Not Completed | 11 | 15 | 16
Not completed — Study Terminated by Sponsor | 8 | 15 | 15
Not completed — Withdrew Consent | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants who were randomized and received at least one dose of study drug.
Groups:
- SIM 75 mg: Blinded Phase: Participants received SIM 75 mg via subcutaneous injection weekly for up to 240 weeks. Open-Label Phase: Participants received SIM 125 mg via subcutaneous injection weekly for up to an additional 240 weeks.
- Total: Total of all reporting groups
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo | Total
Number analyzed (Participants) | 71 | 74 | 74 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8.8) | 53 (9.4) | 53 (8.4) | 53 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 47 | 48 | 138
  Male | 28 | 27 | 26 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 1
  Race: Asian | 1 | 3 | 1 | 5
  Race: Black or African American | 2 | 0 | 1 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Race: White | 66 | 71 | 69 | 206
  Race: Other | 2 | 0 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 9 | 14 | 11 | 34
  Ethnicity: Not Hispanic or Latino | 62 | 60 | 63 | 185
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 6 | 1 | 12
  Belgium | 1 | 1 | 4 | 6
  United States | 51 | 58 | 54 | 163
  Italy | 2 | 2 | 2 | 6
  United Kingdom | 3 | 0 | 5 | 8
  France | 4 | 4 | 4 | 12
  Germany | 3 | 1 | 4 | 8
  Spain | 2 | 2 | 0 | 4
Morphometric Quantitative Collagen (MQC) [Mean (Standard Deviation); unit: percentage of liver collagen] | 7.0 (4.18) | 7.2 (4.62) | 6.7 (3.78) | 7.0 (4.19)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MQC on Liver Biopsy
Time Frame: Baseline to Week 96
Population: Participants in the Full Analysis Set (all enrolled participants who were randomized and received at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of liver collagen
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Number analyzed (Participants) | 46 | 49 | 55
percentage of liver collagen | -3.1 (4.83) | -2.5 (5.11) | -1.9 (4.28)
Statistical Analysis 1: Comparison: SIM 75 mg vs Placebo; A mixed-effect model for repeated measures (MMRM) with an unstructured variance-covariance matrix for each participant was used to calculate a point estimate and a 95% confidence interval (CI) for the treatment difference between each treatment arm and placebo in least squares mean (LSMean) change from baseline in MQC at Week 96. With MMRM setting, all participants with available data from 3 treatment groups with change in MQC at Week 48 and/or Week 96 contributed to the overall model; Test type: Superiority; Difference in LSMeans [SIM - Placebo] = -0.2, 95% CI 2-sided [-1.3 to 1.0]
Statistical Analysis 2: Comparison: SIM 125 mg vs Placebo; An MMRM with an unstructured variance-covariance matrix for each participant was used to calculate a point estimate and a 95% CI for the treatment difference between each treatment arm and placebo in LSMean change from baseline in MQC at Week 96. With MMRM setting, all participants with available data from 3 treatment groups with change in MQC at Week 48 and/or Week 96 contributed to the overall model; Test type: Superiority; Difference in LSMeans [SIM - Placebo] = -0.4, 95% CI 2-sided [-1.5 to 0.8]

2. Primary Outcome: Event Free Survival (EFS) Using Kaplan-Meier
Description: The EFS was the primary clinical efficacy endpoint and was assessed by the time to progression to cirrhosis. Participants were considered to have become cirrhotic if they had a post-baseline biopsy consistent with cirrhosis or developed overt signs and symptoms of cirrhosis. All overt signs and symptoms went through an adjudication process and were confirmed before they were considered for the EFS analysis.
Time Frame: Baseline up to the time of progression to cirrhosis or last dose date (maximum: 240 weeks in the Blinded Phase), which ever occurred first
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- SIM 125 mg: Blinded Phase: Participants received SIM 125 mg subcutaneous injection weekly for up to 240 weeks. Open-Label Phase: Participants received SIM 125 mg subcutaneous injection weekly for up to an additional 240 weeks.
Arm/Group | SIM 75 mg | SIM 125 mg | Placebo
Number analyzed (Participants) | 71 | 74 | 74
months | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [NA to NA] — Data was not estimable as more than 50% of participants were censored. | NA [38.4 to NA] — Data was not estimable as more than 50% of participants were censored.
Statistical Analysis 1: Comparison: SIM 75 mg vs Placebo; Differences in EFS between a given SIM group and placebo were assessed using the log-rank test stratified by the presence or absence of diabetes at baseline; Test type: Superiority; p = 0.73, Stratified log-rank test
Statistical Analysis 2: Comparison: SIM 125 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.85, Stratified log-rank test

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (average exposure: SIM 75 mg= 112.3 weeks, SIM 125 mg= 111.0 weeks, Placebo= 111.3 weeks, Open-label SIM= 51.0 weeks)
Description: Safety Analysis Set included all enrolled participants who were randomized and received at least one dose of study drug and Open-Label Safety Analysis Set included all participants who rolled over into the open-label phase and received at least 1 dose of open-label study drug.
Groups:
- Blinded Phase: SIM 75 mg: Adverse events reported in this group occurred during the Blinded Phase. Participants received SIM 75 mg via subcutaneous injection weekly for up to 240 weeks.
- Blinded Phase: SIM 125 mg: Adverse events reported in this group occurred during the Blinded Phase. Participants received SIM 125 mg via subcutaneous injection weekly for up to 240 weeks.
- Blinded Phase: Placebo: Adverse events reported in this group occurred during the Blinded Phase. Participants received placebo to match SIM via subcutaneous injection weekly for up to 240 weeks.
- Open-Label Phase: SIM 125 mg: All participants who completed the Blinded Phase through the Week 240 visit, or were ongoing at the time the study stopped, or who had progressed cirrhosis of the liver, were offered the opportunity to receive open-label SIM for up to 240 additional weeks. Additionally, participants who developed confirmed progression to cirrhosis prior to completing the Blinded Phase were eligible to roll over into the open-label phase. Adverse events reported in this group occurred during the Open-Label Phase. All participants received fixed-dose open-label SIM 125 mg via subcutaneous injection every week for up to 240 weeks.
Arm/Group | Blinded Phase: SIM 75 mg | Blinded Phase: SIM 125 mg | Blinded Phase: Placebo | Open-Label Phase: SIM 125 mg
Serious Adverse Events (participants affected / at risk) | 17/71 | 17/74 | 14/74 | 11/42
Other Adverse Events (participants affected / at risk) | 65/71 | 69/74 | 72/74 | 29/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase: SIM 75 mg (N=71) | Blinded Phase: SIM 125 mg (N=74) | Blinded Phase: Placebo (N=74) | Open-Label Phase: SIM 125 mg (N=42)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hyperadrenocorticism (Endocrine disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 3 | 2 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Perforation bile duct (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abscess soft tissue (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Phase: SIM 75 mg (N=71) | Blinded Phase: SIM 125 mg (N=74) | Blinded Phase: Placebo (N=74) | Open-Label Phase: SIM 125 mg (N=42)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 4 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 8 | 11 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 4 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 11 | 19 | 17 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Constipation (Gastrointestinal disorders) | 6 | 2 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 19 | 21 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 4 | 1
Nausea (Gastrointestinal disorders) | 16 | 20 | 22 | 5
Vomiting (Gastrointestinal disorders) | 11 | 14 | 10 | 2
Chest pain (General disorders) | 1 | 4 | 6 | 1
Fatigue (General disorders) | 19 | 19 | 24 | 4
Influenza like illness (General disorders) | 2 | 2 | 4 | 0
Injection site bruising (General disorders) | 9 | 3 | 5 | 0
Injection site erythema (General disorders) | 3 | 5 | 0 | 0
Injection site pain (General disorders) | 4 | 1 | 2 | 0
Oedema peripheral (General disorders) | 7 | 3 | 6 | 2
Pain (General disorders) | 3 | 5 | 4 | 1
Pyrexia (General disorders) | 6 | 6 | 5 | 1
Hepatomegaly (Hepatobiliary disorders) | 2 | 1 | 4 | 0
Bronchitis (Infections and infestations) | 16 | 7 | 8 | 1
Cellulitis (Infections and infestations) | 4 | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 4 | 1 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 5 | 1 | 1
Influenza (Infections and infestations) | 8 | 8 | 10 | 2
Localised infection (Infections and infestations) | 4 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 8 | 16 | 1
Sinusitis (Infections and infestations) | 10 | 8 | 14 | 2
Tooth abscess (Infections and infestations) | 6 | 1 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 12 | 10 | 2
Urinary tract infection (Infections and infestations) | 10 | 7 | 14 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 4 | 6 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 2 | 4 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 8 | 6 | 7 | 0
Blood glucose increased (Investigations) | 4 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 5 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 3 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 4 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 4 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 11 | 18 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6 | 20 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 9 | 5 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 8 | 8 | 1
Carpal tunnel syndrome (Nervous system disorders) | 4 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 6 | 7 | 2
Headache (Nervous system disorders) | 12 | 16 | 16 | 2
Anxiety (Psychiatric disorders) | 3 | 5 | 3 | 0
Depression (Psychiatric disorders) | 4 | 5 | 7 | 2
Insomnia (Psychiatric disorders) | 2 | 4 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 10 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 4 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4 | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 7 | 8 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 1
Hypertension (Vascular disorders) | 3 | 5 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years